CLINICAL TRIAL: NCT04878965
Title: Smartwatches to Manage Stress and Anxiety in Residential Settings
Acronym: Smartwatch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 011-2020
Record Dates: First submitted 2021-04-27; First posted 2021-05-10 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Baseline; Technology
Keywords: technology; anxiety; IDD/DD
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: All participants will be provided with a smartwatch to wear.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smartwatch (Other): Individuals receiving the smartwatch
  Interventions: Device: Smartwatch

INTERVENTIONS:
Device: Smartwatch — Smartwatch apparatus to measure strong emotions (e.g., anxiety)

SUMMARY:
The purpose of the study is to conduct a prospective evaluation of a smartwatch technology and an associated application (developed by Awake Labs) in a clinical cohort from Centre for Addiction and Mental Health (CAMH) Adult Neurodevelopmental Services (ANS) and adults with developmental disabilities in the community who have received a watch.

DETAILED DESCRIPTION:
Tools that help predict the onset of anxiety and agitation can not only help a person learn to self-monitor their emotions, but can may also help others feel more efficacious in understanding the internal state of the person they are supporting (especially if not able to communicate), and help them respond in a way that keeps the individual and others safe.

The purpose of the study is to conduct a prospective evaluation of the smartwatch technology with modifications recommended by the researchers (based on a previous retrospective study) in a clinical cohort at CAMH Adult Neurodevelopmental Services (ANS) and in adults with developmental disabilities in the community.

Specifically, this study seeks to evaluate the utility and validity of the smartwatch and associated mobile application as a clinical tool by gathering behavioral data when the applications gives a notification. The person wearing the watch or those in their environment will be asked to report the following in the application after the smartwatch gives a notification: 1) the valence of the emotion of the person wearing the smartwatch, 2) what events were occurring prior to notification (e.g., potential triggers for behaviours that challenge), and 3) what happened after the notification (e.g., how the person or others in their environment responded to the notification).

Results will be used to inform future iterations of the technology and make recommendations for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* individuals with an intellectual and/or developmental disability
* living in the community or receiving services from CAMH ANS department

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Observed/Self-Reported Emotion | 3 months
  What is the person's perceived emotion? The person with the ipod (clinician, support worker) will receive a real-time notification when the smartwatch indicates the individual wearing the watch is experiencing strong emotions. The person with the ipod is to indicate which emotion they are experiencing (e.g., anxiety, happiness)
Observed/Self-Reported Antecedent Events | 3 months
  What was happening before the notification? The person with the ipod (clinician, support worker) will receive a real-time notification when the smartwatch indicates the individual wearing the watch is experiencing strong emotions. The person with the ipod is to indicate what the person who is wearing the smartwatch was doing before immediately before the notification.
Observed/Self-Reported Consequent Events | 3 months
  What happened after the notification?The person with the ipod (clinician, support worker) will receive a real-time notification when the smartwatch indicates the individual wearing the watch is experiencing strong emotions. The person with the ipod is to indicate what happened once they received the notification (e.g., deep breathing)

SECONDARY OUTCOMES:
Accuracy | 3 months
  How accurate is the smartwatch at indicating anxiety? The emotion variable will be used to calculate accuracy of the smartwatch indicating anxiety. This will be calculated by dividing the number of times the smartwatch accurately indicated anxiety (using the number of times the person with the ipod indicated the person wearing the smartwatch was experiencing anxiety) divided by the number of total notifications x100
Incident reports | 2-6 months
  Is there a change in incident reports or the type of incident report before and while wearing the smartwatch. This is a comparison between the total number of incident reports and the types of incident reports before (1-3 months) and while wearing the watch (1-3 months).
PRN | 2-6 months
  Is there a change in the use of PRN before and while wearing the smartwatch. This is a comparison between the total number of PRN delivered before (1-3 months) and while wearing the watch (1-3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Thomson, PhD, BCBA-D, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health - ANS department, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be aggregated before shared with other researchers or published.